CLINICAL TRIAL: NCT07250009
Title: Effect of Silver Diamine Fluoride (SDF) and LED Activation on Residual Caries Activity After Caries Excavation in Class II Primary Molar Cavities"
Brief Title: Effect of Silver Diamine Fluoride and LED Activation on Residual Caries Activity in Class II Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Çanakkale Onsekiz Mart University (Other)
Responsible Party: Principal Investigator, Burak Carıkcıoglu, Assoc. Prof. Dr, Çanakkale Onsekiz Mart University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: CanakkaleOMU3
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SDF Group (Active Comparator): Following caries excavation in Class II primary molar cavities, 38% silver diamine fluoride (SDF) will be applied using a microbrush for 1 minute. Excess material will be gently removed with an air-water spray. No light activation will be performed.
  Interventions: Device: DIAGNOdent measurement
- SDF-LED Group (Experimental): Following caries excavation, 38% SDF will be applied using a microbrush for 1 minute, followed by LED light activation using a blue curing unit (470 nm wavelength, 1000-1200 mW/cm² intensity) for 20 seconds.
  Interventions: Device: DIAGNOdent measurement

INTERVENTIONS:
Device: DIAGNOdent measurement — Residual caries activity will be evaluated with the DIAGNOdent laser fluorescence device (KaVo, Germany) at three time points:
  1. Immediately after caries excavation (D₁ - baseline),
  2. Immediately after SDF application (D₂),
  3. One week after application (D₃). At each time point, DIAGNOdent readings will be recorded three times per site and averaged for analysis.

SUMMARY:
This observational clinical study investigates the effect of silver diamine fluoride (SDF) and its activation with light-emitting diode (LED) on residual caries activity after caries excavation in Class II primary molar cavities. Dental caries in children remains highly prevalent worldwide, and conventional restorative treatments can be difficult in young or uncooperative patients. Minimally invasive approaches such as Atraumatic Restorative Treatment (ART) often leave softened dentin near the pulp, which may remain metabolically active. SDF has been introduced as a simple and effective agent for caries arrest due to its antibacterial and remineralizing effects. However, its optimal application protocol is still under investigation.

Recent studies suggest that LED light exposure after SDF application may enhance its mineralizing effect by accelerating silver ion precipitation, though clinical data remain limited. This study aims to compare the short-term impact of SDF alone and SDF with LED activation on residual caries activity measured quantitatively with the DIAGNOdent laser fluorescence device.

The study will include healthy, cooperative children aged 4-9 years with Class II carious lesions in primary molars. After caries excavation, cavities will receive either SDF alone or SDF followed by 20 seconds of blue LED light (470 nm, 1000-1200 mW/cm²). Residual caries activity will be recorded immediately after application and after one week. The primary outcome is the change in DIAGNOdent readings between groups, while secondary analyses will consider factors such as cavity size, tooth type, and location. The study seeks to clarify whether LED activation enhances the caries-arresting potential of SDF and contributes to evidence-based, minimally invasive strategies in pediatric dentistry.

DETAILED DESCRIPTION:
Dental caries remains one of the most common chronic diseases in childhood, particularly in primary molars where conventional restorative treatment can be difficult due to limited cooperation and treatment-related anxiety. In minimally invasive approaches such as Atraumatic Restorative Treatment (ART), some softened dentin may be intentionally left near the pulp, resulting in residual carious tissue that could remain metabolically active. Preventing this residual activity is critical to ensure lesion arrest and long-term tooth preservation.

Silver diamine fluoride (SDF), especially at 38% concentration, is an established material for caries arrest because of its antibacterial and remineralizing properties. The American Academy of Pediatric Dentistry supports its use as part of minimally invasive dentistry, particularly for young, fearful, or special-needs children. Recent in vitro research suggests that exposure to blue LED light after SDF application may accelerate silver ion precipitation and enhance dentin microhardness, potentially improving the caries-arresting effect. However, clinical data confirming this benefit are limited and inconsistent.

This study aims to evaluate the effect of LED activation on the residual caries activity of SDF-treated Class II primary molar cavities following caries excavation. The research is designed as a non-interventional observational clinical study conducted at the Department of Pediatric Dentistry, Çanakkale Onsekiz Mart University. After caries excavation performed by a pediatric dental specialist, cavities will receive either 38% SDF alone or SDF followed by LED light exposure (470 nm wavelength, 1000-1200 mW/cm² intensity for 20 seconds). All procedures are part of standard clinical practice; researchers will perform only non-invasive fluorescence measurements using the DIAGNOdent device.

Residual caries activity will be recorded at three time points: immediately after excavation (D₁), immediately after SDF or SDF + LED application (D₂), and one week later (D₃). The primary outcome is the change in DIAGNOdent values over time, comparing SDF-only and SDF + LED groups. Secondary outcomes include the influence of cavity size, tooth location, tooth type, and patient sex on these measurements.

Healthy, cooperative children aged 4-9 years with at least one Class II carious lesion in a primary molar that has undergone excavation but not restoration will be included. Children with systemic diseases, allergies to silver, ammonia, or fluoride, pulpal exposure, or infection will be excluded.

By clarifying whether LED activation enhances the effectiveness of SDF, this study aims to contribute clinical evidence for optimizing minimally invasive, child-friendly approaches in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 9 years who apply to the Department of Pediatric Dentistry, Faculty of Dentistry, Çanakkale Onsekiz Mart University.
* Medically healthy children with no systemic or chronic disease.
* Cooperative children who can tolerate clinical procedures and measurements.
* Presence of at least one Class II carious lesion in a primary molar tooth.
* Teeth that have undergone caries excavation by another clinician and received 38% silver diamine fluoride (SDF) application (with or without LED activation).
* Teeth that have not yet been restored after SDF (± LED) treatment.
* Written informed consent obtained from parents or legal guardians through an approved consent form.

Exclusion Criteria:

* Children with systemic or chronic diseases.
* History of allergic reactions or known hypersensitivity to silver, ammonia, or fluoride compounds.
* Uncooperative children or those with insufficient mouth opening during measurement procedures.
* Teeth with pulpal exposure, fistula, abscess, or signs of acute infection.
* Teeth that have previously received any restorative or endodontic treatment.
* Participants who miss the follow-up appointment or whose DIAGNOdent measurements could not be completed.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2025-12-10 (Actual); Primary Completion 2026-01-20 (Actual); Study Completion 2026-01-30 (Actual)

PRIMARY OUTCOMES:
Change in residual caries activity measured by DIAGNOdent laser fluorescence | 1-Immediately after caries excavation (baseline - D₁) 2-Immediately after SDF or SDF + LED application (D₂) 3-One week after treatment (follow-up - D₃)
  Residual caries activity in Class II primary molar cavities will be quantitatively assessed using the DIAGNOdent laser fluorescence device (KaVo, Germany).
  The DIAGNOdent readings (0-99 scale) reflect the fluorescence of carious dentin; higher values indicate greater caries activity. The mean of three consecutive readings per site will be recorded. The primary outcome is the change in DIAGNOdent value from D₁ to D₃, comparing the SDF and SDF + LED groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Canakkale Onsekiz Mart University, Çanakkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided